CLINICAL TRIAL: NCT02115711
Title: A Community Based Approach to Promote Cardiovascular Risk Factor Control in India, Project SEHAT: A Cluster Randomized Controlled Trial
Brief Title: Study of a Community Based Approach to Control Cardiovascular Risk Factors in India
Acronym: SEHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Aditya Khetan, Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 02-14-22
Record Dates: First submitted 2014-04-04; First posted 2014-04-16 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Hypertension; Diabetes; Smoking; Cardiovascular Diseases
Keywords: India; Cardiovascular risk factors; Community health workers; Hypertension; Diabetes; Smoking
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Smoking; Cardiovascular Diseases | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community health worker (Experimental): Home visits by community health worker to deliver the multi-component behavioural intervention targeted at the individual's hypertension, diabetes or smoking.
  Interventions: Behavioral: Community health worker
- Usual care (No Intervention): Patients will receive usual care in the community

INTERVENTIONS:
Behavioral: Community health worker — The intervention is a multi-component one that is tailored to the individual and will target lifestyle changes, health seeking behavior and medication compliance. The CHW, after identifying the cardiovascular risk factors, will give advice about lifestyle interventions and will encourage hypertensives and diabetics to seek a physician. The first phase of the intervention will target hypertension, while the second phase which will be introduced 6 months after the first visit will target diabetes and smoking. The CHW will continue visiting the home of the participants every 2 months to reinforce the previous recommendations, seek to address reasons for non-adherence, address knowledge deficits and encourage physician visits.
  Arms: Community health worker

SUMMARY:
The study is a 2 year community based cluster randomized controlled trial to assess the role that a community health worker led intervention, in concert with physician education, can play in controlling the principal cardiovascular risk factors, i.e. hypertension, tobacco use, diabetes mellitus, physical inactivity and an unhealthy diet. Participants will include around 3600 adults, 35-70 years of age, from the urban community in the town of Dalkhola, Uttar Dinajpur district, West Bengal, India. The hypothesis of the study is that a community health worker based approach can result in increased control of Hypertension, Diabetes and Smoking.

DETAILED DESCRIPTION:
India is currently in the throes of an emerging epidemic of cardiovascular diseases as evidenced by the rising trends in hypertension, smoking and diabetes prevalence observed in the past decade. The country is currently ill equipped to handle this massive problem of chronic diseases. One of the proposed models to address this problem at the primary care level is to expand the pre-existing infrastructure of community health workers that deliver maternal and child health care for screening and management of NCDs. The investigators propose a cluster randomized control study to test the effectiveness of community health workers (CHW) in controlling the three most prevalent cardiovascular risk factors in an integrated manner - hypertension, smoking and diabetes.

The investigators plan to screen around 3600 individuals between the age of 35 and 70 for hypertension, diabetes and smoking from 12 randomly selected clusters in the economically backward urban town of Dalkhola (WB). The screening will be done using house to house visits by CHWs who will administer a questionnaire based on the WHO STEPS survey, measure individual blood pressures and fasting blood glucose. The individuals identified as having atleast one of these risk factors will be eligible for further participation in the study. The clusters will be randomized to either receive the CHW intervention or usual care.

CHWs will be used as the change agents to provide health education, serve as community advocates, and collect data for this study .These CHWs will be chosen from the study population based on a set of criteria through a formal selection panel after consulting with the local leaders and physicians. They will undergo a week of training for the screening process, an additional week for the intervention and finally a refresher course every 6 months. The CHW remunerations will be based on a system of incentives ranging from a minimum of Rs. 12,000 p.a to a maximum of 20,000 p.a.

The intervention is a multi-component one that is tailored to the individual and will target lifestyle changes, health seeking behavior and medication compliance. The CHW intervention will be implemented in a phased manner (2 phases) as is appropriate for multi-component interventions. The CHW after identifying the cardiovascular risk factors will give advice about lifestyle interventions and information about cardiovascular diseases and the benefits of treatment in a one hour session. She will tailor the daily family menu and make appropriate dietary recommendations within the economic context of the family. She will encourage hypertensives and diabetics to seek a physician. The first phase of the intervention will target hypertension, while the second phase which will be introduced 6 months after the first visit will target diabetes and smoking. The CHW will continue visiting the home of the participants every 2 months to reinforce the previous recommendations, seek to address reasons for non-adherence, address knowledge deficits and encourage physician visits. The control group, during their screening visit, will be informed of their problems, given a brief pamphlet and encouraged to seek physician help.

ELIGIBILITY:
Inclusion Criteria:

* All individuals between the ages of 35 and 70 and residing in the area allotted to the CHW will be offered screening.
* Of the screened individuals, those with at least 1 cardiovascular risk factor (either one of Hypertension (BP>140/90), Diabetes (FBG >126) or current daily smoker (self-reported) will be enrolled in the study.

Exclusion Criteria:

* Individuals who are bed-bound because of acute illness, or have a chronic condition that makes them bed-bound.
* Individuals who refuse consent
* Individuals who do not reside in the community and are only visiting, therefore being unlikely to be available for continuous follow up. Individuals who have stayed less than 6 months in the study area, or whose name is not on the voter list of the area will be excluded.
* Individuals who are not able to participate in the intervention due to significant disabilities, such as blindness, deafness or the intellectually disabled.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1242 (Actual)
Dates: Start 2014-04; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Absolute reduction of systolic blood pressure in Hypertensives | 2 years
  Absolute reduction in SBP amongst hypertensives,
  .
Absolute reduction in fasting blood glucose amongst Diabetics | 2 years
  Absolute reduction in fasting blood glucose amongst diabetics
Absolute reduction in average number of cigarettes/bidis smoked per day amongst smokers | 2 years
  Absolute reduction in average number of cigarettes/bidis smoked per day amongst smokers

SECONDARY OUTCOMES:
Absolute mean reduction in DBP amongst hypertensives at end of 2 years | 2 years
Control rates of hypertension at the end of 2 years, control defined as blood pressure less than 140/90 | 2 years
Difference in the Morisky-8 score between the two arms amongst participants who have been prescribed an anti-hypertensive agent at the end of 2 years. | 2 years
Proportion of diabetics whose fasting blood sugars are controlled, defined as fasting blood glucose <126 at the end of 2 years | 2 years
Difference in the Morisky-8 score between the two arms amongst participants who have been prescribed a hypoglycemic agent at the end of 2 years. | 2 years
Proportion of Diabetics who have taken a statin on atleast five of the last seven days as measured at the end of 2 years | 2 years
Proportion of hypertensive smokers who have taken a statin on atleast five of the last seven days as measured at the end of 2 years | 2 years
Proportion of Diabetics who have taken aspirin on atleast five of the last seven days as measured at the end of 2 years | 2 years
Proportion of smokers who have abstained from smoking at the end of 2 years | 2 years
Absolute mean reduction in weight and waist circumference, for those who are overweight or have increased waist size at baseline, at the end of 2 years. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sri Krishna M Mohan, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Rishab Gupta, MD, Principal Investigator — AIIMS, New Delhi, India; Richard Josephson, MS, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Dalkhola, Dalkhola, West Bengal, India

REFERENCES:
- [Derived] Khetan A, Zullo M, Rani A, Gupta R, Purushothaman R, Bajaj NS, Agarwal S, Madan Mohan SK, Josephson R. Effect of a Community Health Worker-Based Approach to Integrated Cardiovascular Risk Factor Control in India: A Cluster Randomized Controlled Trial. Glob Heart. 2019 Dec;14(4):355-365. doi: 10.1016/j.gheart.2019.08.003. Epub 2019 Sep 12. PMID 31523014